CLINICAL TRIAL: NCT01107210
Title: Evaluation of Physical Fitness After Stroke: Evolution and Determinants
Brief Title: Evaluation of Physical Fitness After Stroke
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: National Association for Support to Persons with a Disability NVSG (Unknown); Van Goethem-Brichant foundation (Unknown)
Responsible Party: Ilse Baert, KULeuven
Other Study IDs: ML3617
Record Dates: First submitted 2010-04-13; First posted 2010-04-20 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2010-04

CONDITIONS: Stroke
Keywords: stroke; physical fitness; evolution; determinants
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- stroke patients: 50 patients recruited in the stroke rehabilitation unit in the University Hospital, Leuven, Belgium will be included

SUMMARY:
This study aims to examine the evolution and determinants of physical fitness after stroke.

DETAILED DESCRIPTION:
Stroke is a major cause of chronic severe disability. More than 50% of stroke survivors have residual motor and functional deficits which have an impact on their participation and quality of live (Patel et al, 2006). Limitations on daily functioning may lead to physical inactivity and a sedentary lifestyle. Sustained physical inactivity (deconditioning) induces a reduction in aerobic capacity, which may further increase the risk of cardiovascular diseases in these individuals above that associated with stroke itself. Therefore, improving aerobic capacity may be essential in prevention of secondary diseases due to lack of fitness in the stroke population. Previous studies have also indicated that a critical level of aerobic capacity must be met in order to function independently (Cress et al, 2003). Therefore, in addition to disease prevention, enhancing aerobic capacity in individuals with stroke may also have beneficial effects on promoting functional abilities and independent living. It is also known that a limitation in functional performance is mostly associated with a restriction in social activities (ICIDH-2-model). Clearly, stroke survivors can benefit from counseling on participation in physical activity and exercise training. A recent meta-analysis (Pang et al, 2006) showed that there is good evidence to support the use of aerobic exercise to improve aerobic capacity in individuals with stroke. However, before going on that road, one needs to know more about the level of physical activity and physical fitness in the stroke population.

ELIGIBILITY:
Inclusion Criteria:

1. first-ever stroke as defined by WHO
2. aged < 75 years,
3. able to comprehend simple oral instructions.

Exclusion Criteria:

1. other neurological impairments with permanent damage
2. stroke-like symptoms due to subdural haematoma, tumour, encephalitis or trauma
3. pre-stroke Barthel Index <50
4. unable to perform a maximal exercise test in accordance with absolute contra-indications for exercise testing (ACC/AHA)
5. no informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects with a first ever stroke
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2006-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Evolution of physical fitness after stroke, measured by VO2 peak and OUES. | 1y follow-up
  The criterion standard of cardiorespiratory fitness (VO2max) will be measured during a graded cycle ergometer test. After three minutes of familiarization, the participants will begin to pedal at 10W, with workload increments of 10W/min; they will be instructed to pedal at a comfortable rate between 30 to 60 rpm. Participants will also be monitored with Borg's 16-point Ratings of Perceived Exertion Scale. Maximal effort will be achieved according the ACSM criteria. If no "true" VO2 peak value could be reached, the Oxygen Uptake Efficiency Slope (OUES)will be determined as dependent variable.

SECONDARY OUTCOMES:
Determinants at functional, activity and participation level of physical fitness after stroke | 1y follow-up
  To explore the effect of patient's demographic characteristics and initial stroke severity on the evolution of cardiorepiratory fitness, following independent variables will be used: age, gender, BMI, pre-stroke activity level, type of stroke, NIHSS, TIS, RMA-GF, FAC, BI and MMSE. Patient's functional level (lower limb strength), activity level (TIS, RMA-GF, FAC, BI, NEADL, timed 10m test), participation level (MMSE, BDI-II, SIP 3.0, MRS); patient's body composition (BMI, skinfolds); and use of health services will be assess to identify determinants of cardiorespiratory fitness.

CONTACTS AND LOCATIONS:
Overall Officials: Ilse Baert, Msc, PT, Principal Investigator — KU-Leuven, Faculty of Movement and Rehabilitation Sciences; Yves Vanlandewijck, PhD, Study Chair — KU-Leuven, Faculty of Movement and Rehabilitation Sciences; Daniel Daly, PhD, Study Chair — KU-Leuven, Faculty of Movement and Rehabilitation Sciences; Hilde Feys, PhD, Study Chair — KU-Leuven, Faculty of Movement and Rehabilitation Sciences
Locations (1):
- University Hospital Leuven, Rehabilitation Centre Pellenberg, Pellenberg, Belgium